CLINICAL TRIAL: NCT00917436
Title: Thiocolchicoside Injection and Capsule in Treatment of Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: L_9826
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — thiocolchicoside

INTERVENTIONS:
Drug: Thiocolchicoside

SUMMARY:
To assess two regimens of thiocolchicoside injection and capsule in combination with either diclofenac or ibuprofen in patients with acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute low back pain of recent onset (less than 7 days) and defined by spontaneous pain intensity at rest more than or equal to 50mm of the visual analog scale.
* Presence of lumbar muscular contracture

Exclusion Criteria:

* Acute low back pain due to vertebral collapse or neoplastic, inflammatory (ankylosing spondylitis), or infective origins
* Patients with psychiatric or mental diseases, or unable to follow the requests of the protocol
* Renal failure (serum creatinine > 160 µmol/l or > 1.80 mg/dl) and/or severe hepatic dysfunction (alanine aminotransferase and/or aspartate aminotransferase and/or total bilirubin > 2 Upper normal limit).
* Positive history of cerebro-vascular accidents or myocardial infarction in the six months prior the inclusion.
* Severe heart failure.
* Myopathy / myasthenia.
* Patients treated during two days prior to inclusion with steroidal agents.
* Known or suspected hypersensitivity to thiocolchicoside.
* Known or suspected hypersensitivity to nonsteroidal anti-inflammatory drugs
* History of active peptic ulcer or gastro intestinal bleeding.
* History of nonsteroidal anti-inflammatory drugs induced allergic asthma.
* Concomitant treatment with 2-agonists (i.e. clonidine).
* Pregnant or breast feeding women.
* Females of child bearing potential, not taking adequate contraception.
* Patients with history of alcohol, drugs or narcotics abuse.
* Previous inclusion in this study or in another study in the past 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Pain score evaluated by patient-rated visual analog scale: the levels of spontaneous pain is indicated by the patient by means of a 10 centimetre non-graduated scale, in which the patient could estimate the intensity of pain | During patient visits: day 1, day 3 and day 5 to 10

SECONDARY OUTCOMES:
Mobility Hand-to-floor distance is evaluated by a simple graduated bar (0 value at floor). | During patient visits: day 1, day 3 and day 5 to 10
Disability Questionnaire (Roland Morris) | During patient visits: day 1, day 3 and day 5 to 10
Physician rated Clinical Global Impression Scale | During patient visits: day 1, day 3 and day 5 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Manish MISTRY, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Mumbai, India